CLINICAL TRIAL: NCT00101621
Title: A Randomized, Double-Blind, Placebo Controlled, Multi-Center, Pilot Study to Evaluate the Safety and Analgesic Activity of M40403 Co-Administered With an Opioid Agent in a Cancer Pain Model
Brief Title: Pilot Study to Evaluate the Safety and Analgesic Activity of M40403 Co-Administered With an Opioid Agent for Cancer Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: MetaPhore Pharmaceuticals (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: U10-04-02-007
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2006-02-09 (Estimated); Status verified 2006-02

CONDITIONS: Cancer; Pain
Keywords: cancer; pain; Cancers, Pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — imisopasem manganese

INTERVENTIONS:
Drug: M40403

SUMMARY:
M40403 was found to be effective in reducing pain in animal models and in clinical studies of subjects who were experiencing pain after dental surgery. The proposed study is designed to investigate the efficacy and safety of M40403 when co-administered with an opioid in subjects with pain due to cancer.

DETAILED DESCRIPTION:
The proposed study is designed to investigate the efficacy, safety, and pharmacokinetics of M40403 in subjects with pain related to cancer. Because the effects of M40403 have not been previously investigated in subjects with cancer-related pain, the safety of single doses of 0.0625, 0.125, and 0.25 mg/kg of M40403 will be evaluated in an open label phase of the study. These doses of M40403 are similar to doses that were used in subjects who were experiencing pain in prior clinical studies with M40403.

ELIGIBILITY:
Inclusion Criteria:

* Has somatic or visceral pain due to solid tumor cancers (adrenal, basal cell, and breast cancers; transitional cell carcinoma of the bladder or uroepithelium; cholangiocarcinoma; small intestine/colon/rectal cancers; adenocarcinoma, esophageal/gastric cancers; hepatocellular, ovarian, pancreatic, and prostate cancers; bony/soft tissue sarcomas; small cell lung cancer; non small cell lung cancer; and adenocarcinomas of unknown primary origin).
* Has moderate to severe pain as measured by the Pain Intensity Assessment (categorical scale), and a pain intensity measurement of greater than or equal to 40 mm by visual analog scale (VAS) prior to the morning dose of pain medication.
* Stable chronic cancer pain as evidenced by a stable, scheduled opioid regimen over 7 days prior to treatment with study medication and fewer than 3 rescue doses per day averaged over the 3 days prior to treatment with study medication.
* Currently taking morphine, hydromorphone, oxycodone or an oxycodone/acetaminophen combination for the treatment of cancer pain.
* Age 18 or older.
* Performance status of 0 to 2 by Eastern Cooperative Oncology Group (ECOG) scale.
* If taking concomitant medication, subject has been on a steady regimen for the past 2 weeks.
* For female subjects: 2 years postmenopausal or currently using effective contraception, and not lactating; negative urine pregnancy test within 24 hours of randomization.
* Weight of 40 to 90 kg and body mass index (BMI) of 18 to 32 during a 1-week period prior to treatment.
* Able to remain at facility allowing completion of pain and safety assessments for at least 8 hours after receiving study medication.

Exclusion Criteria:

* Has any significant medical disease other than malignancy that, in the Investigator's opinion, may interfere with study participation or completion of the study.
* Has a history of chronic analgesic or tranquilizer use (except for the subject's current pain medication [morphine, hydromorphone, and oxycodone, or an oxycodone/acetaminophen combination]) or known substance abuse within 90 days prior to the screening visit. Other drugs with analgesic properties, including nonsteroidal anti-inflammatory drugs, corticosteroids, tricyclic antidepressants, anticonvulsants, antiarrhythmics, bisphosphonates or gabapentinoids will not be initiated during the study. Patients receiving stable doses of these agents for pain management or other indications for >1 week prior to the screening visit may continue treatment with these provided that the dose remains constant during the study.
* Is unwilling to abstain from alcohol from at least 8 hours prior to dosing with study medication until time of discharge from the study unit.
* Has received or anticipates receiving any vitamin and mineral supplements from 24 hours prior to dosing until time of discharge from the study unit.
* Has received any investigational medication within 30 days prior to administration of study medication or is scheduled to receive an investigational drug other than study drug during the course of this study.
* Has clinically significant hypersensitivity to morphine, oxycodone, hydromorphone, other opioids, nonsteroidal anti-inflammatory drugs (NSAIDs), or acetaminophen.
* Has a laboratory abnormality that, in the opinion of the Investigator, would contraindicate study participation, including aspartate aminotransferase (AST), alanine aminotransferase (ALT), or blood urea nitrogen (BUN) levels greater than or equal to 1.5 times the upper limit of normal (ULN) or creatinine level greater than ULN at the screening evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-08; Study Completion 2005-08

PRIMARY OUTCOMES:
To evaluate the safety and analgesic activity of a single dose of 0.25 mg/kg (or the highest tolerated dose from the open-label phase) of M40403 co-administered with current pain medication in subjects experiencing moderate to severe pain.

SECONDARY OUTCOMES:
To evaluate safety and analgesic activity of ascending, single doses of M40403 (0.0625, 0.125, and 0.25mg/kg) co-administered with current pain medication and to assess the pharmacokinetic parameters of a single dose of M40403.

REFERENCES:
- See also: Visit Metaphore Pharmaceuticals website to learn more about the company, its products and clinical trials. — http://www.metaphore.com